CLINICAL TRIAL: NCT02034292
Title: Phase I Study to Assess the Safety of APD-791 When Co-administered With Aspirin
Brief Title: Safety Study of APD-791 With Aspirin and/or Clopidogrel
Acronym: TG1C
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: ID-TG1C-1301
Record Dates: First submitted 2013-12-12; First posted 2014-01-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Aspirin; APD791

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 10mg MD (Experimental): APD791 10mg Multiple dose and
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 20mg MD (Experimental): APD791 20mg Multiple dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 40mg MD (Experimental): APD791 40mg Multiple dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 60mg MD (Experimental): APD791 60mg Multiple dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- Placebo MD (Placebo Comparator): Placebo for Multiple dose group
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 120mg SD (Experimental): APD791 120mg Single dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 240mg SD (Experimental): APD791 240mg Single dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- 320mg SD (Experimental): APD791 320mg Single dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: APD791
- Placebo SD (Placebo Comparator): Placebo for Single dose
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel
Drug: Aspirin
Drug: APD791
  Arms: 10mg MD; 120mg SD; 20mg MD; 240mg SD; 320mg SD; 40mg MD; 60mg MD; Placebo MD
Drug: Placebo
  Arms: Placebo SD

SUMMARY:
Evaluating safety and PK parameter of APD-791 when co-administered with aspirin and clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

1. a healthy adult between 20 and 45 years old at the time of visit for screening
2. a person who is able to give written consent
3. a person between 50 and 85 kg at the time of visit for screening
4. a woman who is negative on a serum hCG test at the time of visit and the day before a trial, and who is not nursing
5. a woman who agrees on double contraception, medically approved, from the time of visit for screening to 90 days after the last administration of a clinical trial drug, or who had a contraceptive operation no later than 120 days before visit for screening, or who is menopausal
6. a man who had a contraceptive operation no later than 120 days before visit for screening, or who agrees on double contraception, medically approved, from the time of visit for screening to 90 days after the last administration of a clinical trial drug, and also agree not to donate sperm
7. a person more than hemoglobin 12 g/dL at the time of screening (a woman more than hemoglobin 11 g/dL)
8. a person whose vital signs were in the normal range at the time of visit for screening, or who is medically determined not to be clinically significant by an investigator
9. a person who voluntarily decides to participate in this clinical trial and gives written consent on strict clinical trial compliance
10. a person whose blood can be collected during a study period with visit for monitoring

Exclusion Criteria:

1. a person with the medical history of gastric ulcer, duodenal ulcer or esophageal ulcer within 90 days from the time of visit for screening
2. a person with the medical history of gastrointestinal diseases(e.g. Crohn's disease, ulcerative colitis, etc.) or surgery(excluding uncomplicated appendectomy or herniotomy) affecting the absorption of a clinical trial drug
3. a person with the medical history of blood coagulation disorder or hemorrhagic diseases, or with clinically significant abnormal findings decided by a investigator on blood coagulation test at the time of screening
4. a woman with the medical history of dysfunctional uterine bleeding within a year from the time of visit for screening
5. a person with the medical history of epilepsy or convulsion
6. a person with the medical history of internal organ transplant
7. a person expected to be hard to complete a clinical trial because of surgery or medical procedures planned within a clinical trial period
8. a person with the medical history of clinically significant new diseases within 30 days from the time of visit for screening according to investigator's decision
9. a person with hypersensitivity reaction to a drug or gelatin, or the medical history of clinically significant hypersensitivity reaction
10. a person with the history of drug abuse, or with a positive reaction to a drug possible to be abused on urine drug screening
11. a person with the medical history of alcohol abuse within two years from the time of visit for screening
12. a person who is a smoker, or with a positive reaction on a urine nicotine test conducted at the time of visit for screening
13. a person who donated whole blood within 60 days or constituents of blood within 30 days, or received a blood transfusion within 30 days from the time of visit for screening
14. a person taking other clinical trial drugs within 90 days from the time of visit for screening
15. a person taking a prescription drug within 30 days, or a contraindicated drug or oriental medicine within 14 days from the time of visit for screening
16. a person with a positive reaction to a serum test(hepatitis B test, hepatitis C test, HIV test, syphilis test)
17. a person with hepatic enzymes(AST, ALT) more than 2.5 times of the reference upper limit(UNL) or total bilirubin more than 1.5 times of the reference upper limit(UNL) or creatinine more than 1.25 times of the reference upper limit(UNL)
18. a person expected to be hard to complete a clinical trial due to physical or mental status according to investigator's medical decision at the time of visit for screening
19. a person decided to be inappropriate to participate in this clinical trial according to investigator's medical decision on the result of laboratory tests, such as complete blood cell count, general chemical test, clinicochemical urinalysis, and physical examination, vital signs, ECG, other tests excluding exclusion criteria 17 items conducted before subject selection for a clinical trial

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety of APD791 when orally co-administered with Aspirin and Clopidogrel in healthy subjects | safety review will be conducted at every end of dosing (about every 2 or 3 weeks)
  Adverse reaction monitoring for subjective or objective symptoms Physical examination Vital signs 12-electrode ECG Laboratory tests

SECONDARY OUTCOMES:
Pharmacokinetic characteristic evaluation variable | After last patient last visit. About 8month later since start of the study.
  Non-compartmental analysis is conducted by using APD791 and its metabolite, M1 and M2 and the following pharmacokinetic evaluation variables are calculated.
  Cmax0-12, Cmax,ss (Day 7 only), Cmin,ss (Day 7 only), tmax0-12, tmax,ss (Day 7 only), λz, t1/2β, AUC0-12 (Day 1 only), AUCinf, Accumulation index, CL/F, MRT, Vz/F
Pharmacodynamic characteristic evaluation variable | Day1, Day4, Day7 of every dose for mutiple dose group and first day for single dose group.
  Pharmacodynam1) % inhibition of serotonin-stimulated platelet aggregation 2) Change in % inhibition of serotonin-stimulated platelet aggregation 3) % inhibition of TRAP-induced platelet aggregation ic characteristic evaluation variable